CLINICAL TRIAL: NCT02052570
Title: School Reintegration After Pediatric Hematopoietic Stem Cell Transplant: Experiences of Children, Parents, Teachers and Providers
Brief Title: School Reintegration After Pediatric Hematopoietic Stem Cell Transplant
Status: Withdrawn | Type: Observational
Why Stopped: Unable to meet all criteria as outlined for participants
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00047417
Record Dates: First submitted 2014-01-27; First posted 2014-02-03 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Unspecified Complication of Bone Marrow Transplant
Keywords: School Reentry after pediatric HSCT

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Children post-HSCT: Children post-HSCT age 10-16 yrs of age who had allogeneic transplant who are within 5 years of transplant and returned to school in past 12-24 months after previously attending school pre-transplant
- Parents of children post-HSCT: Parents of children post-HSCT (children in focus group) will participate in focus group with other parents to discuss the challenges and successes of their child returning to school following HSCT.
- Teachers of children post-HSCT: Teachers of children post- HSCT (children in focus group) will participate in focus group with other teachers to discuss the challenges and successes of children returning to school post HSCT
- PBMT provider of child post-HSCT: PBMT provider of child-post HSCT (child in focus group) will participate in in focus group with other PBMT providers to discuss the successes and challenges of coordinating school reentry in child post-HSCT

SUMMARY:
This is a qualitative study that will explore the experiences of school reentry following Hematopoietic Stem Cell Transplant (HSCT) in children ages 10-16 years of age, their parents, teachers and primary PBMT(Pediatric Bone Marrow Transplant) providers. This study will involve four focus groups: children post -transplant, parents, teachers and PBMT providers in an effort to understand the successes and challenges of returning to school following HSCT.

DETAILED DESCRIPTION:
This is a qualitative descriptive study using purposive sampling to form the four focus groups to encourage diversity in diagnosis (immunodeficiency, malignancy, bone marrow failure and inherited metabolic diseases), age and location. Each group will participate via conference call due to difference in location. There will be semi-structured questions for each group but also allow flexibility by participants themselves.

ELIGIBILITY:
Inclusion Criteria:

* Children transplanted in the PBMT program at DUMC in the past 5 years for allogeneic HSCT to include diagnoses for malignancy, immunodeficiency, bone marrow failure and inherited metabolic disease. They must have previously attended school prior to transplant

Exclusion Criteria:

* Autologous transplants
* Significant developmental delays that would impair ability to communicate
* Inability to get full team (child, parent, teacher, provider) to participate
* Non-English speaking

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children transplanted in the PBMT (Pediatric Bone Marrow Transplant) program at DUMC (Duke University Medical Center) in the past 5 years for allogeneic HSCT to include diagnoses for malignancy, immunodeficiency, bone marrow failure and inherited metabolic disease. They must have previously attended school prior to transplant.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Psychosocial issues | 90 minutes
  Psychosocial issues related to school reentry following pediatric hematopoietic stem cell transplant (HSCT) as gathered from children's, parent's, teacher's and health care provider's perspectives as obtained during focus group discussions.
Cultural and environmental issues | 90 minutes
  Cultural and environmental issues (ie location, resources) issues related to school reentry following pediatric hematopoietic stem cell transplant (HSCT) gathered from the children's, parent's, teacher's and health care provider's perspectives as obtained during focus group discussions.

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Wood, MN, Principal Investigator — DUMC
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States